CLINICAL TRIAL: NCT07319598
Title: A Randomized, Double-Blind, Placebo-Controlled Clinical Study to Evaluate the Efficacy and Safety of Tetrandrine Tablets in Treating Interstitial Lung Disease Related to Connective Tissue Disease
Brief Title: A Study to Test Tetrandrine Tablets for Connective Tissue Disease-Related Lung Disease
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: V1.5/2024.11.08
Record Dates: First submitted 2025-08-27; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-08

CONDITIONS: Interstitial Lung Disease (ILD); Connective Tissue Disease-associated Interstitial Lung Disease
Keywords: Tetrandrine; Connective Tissue Disease; Interstitial Lung Disease; Pulmonary Function; Inflammatory Markers
MeSH Terms: conditions — Lung Diseases, Interstitial; Connective Tissue Diseases | interventions — tetrandrine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tetrandrine Group (Experimental): Participants receive tetrandrine tablets (60 mg, three times daily) for 24 weeks, along with standard treatment (glucocorticoids and immunosuppressants).
  Interventions: Drug: Tetrandrine Tablets
- Placebo Group (Placebo Comparator): Participants receive placebo tablets (mimicking tetrandrine, three times daily) for 24 weeks, along with standard treatment (glucocorticoids and immunosuppressants).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tetrandrine Tablets — 60 mg (3 tablets, 20 mg each), orally three times daily (TID) for 24 weeks, with glucocorticoids and immunosuppressants
  Arms: Tetrandrine Group
Drug: Placebo — Placebo tablets mimicking tetrandrine, 3 tablets TID, orally for 24 weeks, with glucocorticoids and immunosuppressants
  Arms: Placebo Group

SUMMARY:
This study evaluates the efficacy and safety of tetrandrine tablets (60 mg, three times daily) compared to placebo in adult patients with connective tissue disease-related interstitial lung disease. Patients receive standard treatment (glucocorticoids and immunosuppressants) alongside the study drug or placebo for 24 weeks. The study measures changes in lung function, inflammatory markers, lung imaging, quality of life, and safety outcomes.

DETAILED DESCRIPTION:
This multicenter, randomized, double-blind, placebo-controlled study enrolls 100 adults with connective tissue disease-related interstitial lung disease. Patients are randomized 1:1 to receive tetrandrine tablets (60 mg TID) or placebo for 24 weeks, alongside standard treatment. The primary outcome is the change in forced vital capacity (FVC) at 24 weeks. Secondary outcomes include changes in serum inflammatory markers (TGF-β1, KL6, TNF-α, IL-6), lung HRCT scores, other Lung function parameters (TLC, VC, DLCO, PaO2), St. George's Respiratory Questionnaire (SGRQ) score, safety parameters, and all-cause mortality. Visits occur at weeks 4, 8, 12, and 24 for efficacy and safety assessments.

ELIGIBILITY:
Inclusion Criteria:

* Patients who voluntarily participate and sign the informed consent form
* Male or female patients aged 18-80 years (inclusive)
* Patients meeting the diagnostic criteria for connective tissue disease-related interstitial lung disease per the 2018 Chinese Expert Consensus at screening
* FVC ≥40% of predicted value at screening
* Fertile male or female patients must agree to use effective contraception from signing informed consent until 3 months after the last study drug dose (Exemptions: postmenopausal women >50 years with amenorrhea for >1 year, or surgically sterilized women)
* Patients on stable doses of prednisone (≤20 mg/day or equivalent) or immunosuppressants for at least 4 weeks prior to study entry, with dose adjustments not exceeding this during the double-blind period

Exclusion Criteria:

* Treatment with tetrandrine or other antifibrotic drugs within 1 month before screening
* Diabetes with fasting blood glucose greater than 11.1 mmol per L
* Resting arterial oxygen partial pressure less than 50 mmHg
* Active peptic ulcers or bleeding disorders
* Tumors with expected survival less than 1 year
* Active pulmonary tuberculosis
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) 5 times the upper limit of normal (ULN) or higher, or ALT or AST 3 times ULN or higher with total bilirubin 2 times ULN or higher
* Creatinine clearance less than 30 mL per min (per Cockcroft-Gault formula) or patients receiving dialysis
* Known allergy to tetrandrine or its excipients
* Severe psychological, mental, cognitive, or intellectual impairments that may affect compliance
* Pregnant or breastfeeding women, or those planning pregnancy within 3 months after the last study drug dose
* Participation in another clinical trial within 3 months before screening
* Patients deemed unsuitable for the study by the investigator
* Clinically significant environmental exposure history that may cause pulmonary fibrosis (e.g., amiodarone, asbestos, beryllium, radiation)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-11-02 (Actual); Primary Completion 2026-10-15 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Change in Forced Vital Capacity (FVC) | Baseline to 24 weeks
  Change in forced vital capacity (FVC) expressed in liters (L) of predicted normal value, measured using a pulmonary function testing device in accordance with ATS/ERS standards at a central facility. Units: Absolute value（L）

SECONDARY OUTCOMES:
Change in Serum Transforming Growth Factor Beta 1 (TGF-β1) Level | Baseline to 24 weeks
  Serum TGF-β1 levels measured via fully automated analyzer. Units: ng/mL
Change in Serum Krebs von den Lungen-6 (KL6) Level | Baseline to 24 weeks
  Serum KL6 levels measured via fully automated analyzer. Units: U/mL
Change in Serum Tumor Necrosis Factor Alpha (TNF-α) Level | Baseline to 24 weeks
  Serum TNF-α levels measured via fully automated analyzer. Units: pg/mL
Change in Serum Interleukin-6 (IL-6) Level | Baseline to 24 weeks
  Serum IL-6 levels measured via fully automated analyzer. Units: pg/mL
Change in Semi-Quantitative High-Resolution Computed Tomography (HRCT) Score | Baseline to 24 weeks
  Semi-quantitative scoring of HRCT patterns (reticulation, ground-glass opacity, patchy/consolidation, honeycombing) across 6 predefined lung layers. Each pattern scored 0 (absent) to 4 (>75% involvement); total score summed (maximum 96). Higher scores indicate worse outcome (greater lung involvement). Units: Score (0-96)
Change in Total Lung Capacity (TLC) | Baseline to 24 weeks
  TLC measured via body plethysmography (ATS/ERS standards) at central facility. Units: Absolute value（L）
Change in Vital Capacity (VC) | Baseline to 24 weeks
  VC measured via spirometry (ATS/ERS standards) at central facility. Units: Absolute value（L）
Change in Diffusing Capacity of the Lung for Carbon Monoxide (DLCO) | Units: Absolute value（L）
  Single-breath DLCO (hemoglobin-corrected) measured via ATS/ERS standards at central facility.
Change in Arterial Partial Pressure of Oxygen (PaO2) | Baseline to 24 weeks
  PaO2 from arterial blood gas (at rest, room air). Units: mmHg
Change in St. George's Respiratory Questionnaire (SGRQ) Total Score | Baseline to 24 weeks
  Change in total score from Chinese-validated SGRQ (self-administered, 3-month recall), assessing respiratory health-related quality of life across Symptoms, Activity, and Impacts domains (weighted). Scores range from 0 (no impairment/best quality of life) to 100 (maximum impairment/worst quality of life). Higher scores indicate worse outcome. Units: Score (0-100)
Number of Participants with Treatment-Related Adverse Events as Assessed by CTCAE v5.0 | Baseline to 24 weeks
  Incidence of treatment-related adverse events (any untoward event post-randomization), graded by CTCAE v5.0 (coded via MedDRA). Includes abnormalities in hematology, chemistry, urinalysis, liver/kidney function. Units: Number of cases
Number of Participants with Treatment-Emergent Serious Adverse Events | Baseline to 24 weeks
  Incidence of serious adverse events as assessed by CTCAE v5.0. Units: Number of cases
Number of Participants with Clinically Significant Abnormalities in Electrocardiogram (ECG) | Baseline to 24 weeks
  Incidence of clinically significant ECG abnormalities (e.g., QTc prolongation) from 12-lead ECGs. Units: Number of cases
Number of Participants with All-Cause Mortality | Baseline to 24 weeks
  Number and percentage of participants who died from any cause during the study period (all-cause mortality), ascertained via follow-up and vital status checks. Units: Number of cases

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, China